CLINICAL TRIAL: NCT06682520
Title: Evaluation of a Health System Integrated Model for Postpartum Education and Support in Rural Populations - NEST-Rural
Brief Title: Evaluation of a Health System Integrated Model for Postpartum Education and Support in Rural Populations
Acronym: NEST-Rural
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00113575
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Health Care Utilization
Keywords: Remote blood pressure monitoring; Postpartum Nurse home visiting; Postpartum Health Care Services; Postpartum Hospital Program Service Model; Maternal Health; Newborn Health
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Randomization to one of two study arms: Postpartum Standard of Care (Control arm). Postpartum NEST-Rural Program Service model (Experimental arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postpartum NEST-Rural Program Group (Experimental): Postpartum women randomized to this group will receive the usual postpartum care from an Obstetrics provider and the following NEST-Rural Program:
  * Information about services and resources available in your community
  * A blood pressure monitor.
  * Access to the Babyscripts smartphone app.
  * A nurse visit(s) at home or via telehealth.
  * A visit(s) from a Family Outreach Specialist, if needed.
  * A follow-up phone call from a Coordinator in about 6 weeks
  Interventions: Other: Postpartum NEST-Rural Program (Hospital based service model)
- Postpartum Usual Care Group (No Intervention): Postpartum women randomized to this group will receive the usual postpartum care from an Obstetrics provider and the following:
  * Information about services and resources available in your community
  * A follow-up phone call from a Coordinator in about 6 weeks

INTERVENTIONS:
Other: Postpartum NEST-Rural Program (Hospital based service model) — NEST-Rural services will include 3-5 nurse encounters and, if indicated, up to 3 social work encounters with mothers and their infants in the postpartum period, postpartum remote blood pressure monitoring, breastfeeding support, infant weight checks, linking mothers and infants to needed social, behavioral, and health-related resources, and integration of service delivery with healthcare providers.
  Arms: Postpartum NEST-Rural Program Group

SUMMARY:
This study was designed to evaluate the implementation of the Nurse Education and Support Team (NEST) Program for postpartum women who reside in 5 rural counties in North Carolina. Overarching Hypothesis: Mothers and infants residing in rural communities, randomized to the NEST-Rural care model over the 3-year course of the project will: 1. Receive more coordinated care for addressing social, mental and physical health needs. 2. Experience fewer postpartum hospital readmissions and decreased utilization of emergency departments (ED) for healthcare. 3. Experience higher adherence to American College of Obstetricians and Gynecologists (ACOG) and American Academy of Pediatrics (AAP) guidelines for preventive care, including recently updated ongoing postpartum care, serial well-child visits and vaccinations compared to those assigned to usual care. This group will be compared to those assigned to usual care,

DETAILED DESCRIPTION:
This is a Randomized Control Trial (RCT) designed study evaluating the implementation of the Nurse Education and Support Team (NEST) Program for postpartum women who reside in 5 rural counties (Davie, Davidson, Yadkin, Wilkes and Stokes counties) in North Carolina. The study cohort will be for all mothers residing in these rural counties and delivering their infant(s) in the Atrium Health Wake Forest Baptist Birth Center. It is anticipated that 1,300 mother-infant dyads will be enrolled and randomized to either usual care [visit 4-6 weeks postpartum] (~650) or NEST-Rural care (~650).

The NEST model is unique in that it supports both maternal and infant health, with an emphasis on using strategies aligned with evidence-based guidelines for postpartum and infant healthcare. Another important feature of NEST is integration of service delivery in the healthcare system. This integration facilitates reaching mother-infant dyads and bi-directional communication with the mother's and infant's healthcare providers to enable appropriate, timely healthcare. For example, as part of NEST, mothers are discharged from the hospital with a remote blood pressure monitor. Blood pressures are transmitted to a service hub through an app that is downloaded onto her phone prior to hospital discharge. The hub alerts the healthcare team, which follows-up with her to determine appropriate care.

Randomization to NEST-Rural services will include 3-5 nurse encounters with mothers and their infants in the postpartum period, postpartum remote blood pressure monitoring, breastfeeding support, infant weight checks, linking mothers and infants to needed social, behavioral, and health-related resources, and integration of service delivery with healthcare providers. Services will initiate in the postpartum hospital unit, with a NEST Coordinator introducing the program and identifying and making referrals and/or providing resources for emergent needs (e.g. pack-n-play, diapers), and offering and scheduling a follow-up nurse visit (home or telehealth-based, depending on needs) 2-3 weeks postpartum. Up to two additional nurse and/or social worker home/virtual visits will be provided, depending on the family's needs. At six weeks postpartum, the NEST Coordinator will contact the family to inquire whether any referrals were made and assess for continuing gaps in support. Following nurse encounters, a note will be sent to the mother's and infant's healthcare providers. If acute concerns are identified, the nurse will contact the provider immediately for additional care.

ELIGIBILITY:
Inclusion Criteria:

1. Women that deliver an infant(s) at The Birth Center at Atrium Health Wake Forest Baptist and currently reside in Davidson, Davie, Stokes, Wilkes or Yadkin County in North Carolina
2. Women that delivered an infant(s) at home, were transported to Atrium Health Wake Forest Baptist and received postpartum care at The Birth Center and currently reside in Davidson, Davie, Stokes, Wilkes or Yadkin County in North Carolina
3. Ages 18 years or older

Exclusion Criteria:

1. Women that delivered an infant(s) and did not receive postpartum care at The Birth Center at Atrium Health Wake Forest Baptist.
2. Women that currently reside outside of Davidson, Davie, Stokes, Wilkes or Yadkin County in North Carolina
3. Under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Median number of hospital readmissions - Maternal | Baseline through 30 days postpartum
  Number of hospital readmissions in the 4th trimester
Median number of hospital readmissions - Maternal | Baseline through 90 days postpartum
  Number of hospital readmissions in the 4th trimester
Median number of encounters for urgent or emergent care - Maternal | Baseline through 30 days postpartum
  Number of visits to Urgent Care or the Emergency Room in the 4th trimester
Median number of encounters for urgent or emergent care - Maternal | Baseline through 90 days postpartum
  To determine number of visits to Urgent Care or the Emergency Room in the 4th trimester
Proportion of women that attend recommended postpartum visits | Baseline through 90 days postpartum
  Percentage of women that attended recommended visits to their obstetrician after delivery.
Median number of hospital readmissions - Infant | Baseline through 30 days postpartum
  Number of hospital readmissions after birth following hospital discharge.
Median number of hospital readmissions - Infant | Baseline through 90 days postpartum
  Number of hospital readmissions after birth following hospital discharge.
Median number of encounters for urgent or emergent care - Infant | Baseline through 30 days postpartum
  Number of visits to Urgent Care or the Emergency Room following hospital discharge.
Median number of encounters for urgent or emergent care - Infant | Baseline through 90 days postpartum
  Number of visits to Urgent Care or the Emergency Room following hospital discharge.
Proportion of infants receiving a visit with an ambulatory care provider | Baseline through 21 days postpartum
  Percentage of infants that attended recommended visits to their pediatric care provider within 21 days following hospital discharge
Proportion of infants that received >/= 4 well-child care visits with an ambulatory care provider | Baseline through 274 days postpartum
  Percentage of infants that attended recommended visits to their pediatric care provider within the first 9 months following hospital discharge

SECONDARY OUTCOMES:
Median number of days with >/= 1 remote blood pressure obtained - Maternal | Baseline through 21 days postpartum
  Number of days that patients checked and remotely reported their blood pressure readings following hospital discharge.
Proportion of women with a diagnosis of hypertensive disorders of pregnancy with at least one blood pressure obtained | Baseline through 10 days postpartum
  Percentage of women diagnosed with hypertensive disorders that checked and remotely reported at least one blood pressure reading.
Proportion of women with preeclampsia with severe features with at least one blood pressure obtained | Baseline through 3 days postpartum
  Percentage of women with preeclampsia with severe features checked and remotely reported at least one blood pressure reading.
Proportion of women exceeding 3 days length of stay in hospital after delivery | Baseline through date of hospital discharge
  Percentage of women that remain hospitalized for more than 3 days following delivery.
Median length of stay for hospital readmissions after delivery | Baseline through 90 days postpartum
  Number of days mothers are readmitted and remain hospitalized after delivery.
Proportion of women that attend a follow-up encounter with their primary care physician | Baseline through 365 days postpartum
  Percentage of women that have a follow-up visit with their primary care physician within the first year after giving birth.
Proportion of women who receive a nurse home visit | Baseline through 30 days postpartum
  Percentage of women who receive a nurse home visit within 30 days of discharge
Proportion of women eligible for an in-person home visit that received the in-person nurse visit | Baseline through 30 days postpartum
  Percentage of women eligible for an in-person nurse home visit that received the in-person home visit.
Proportion of women eligible for an in-person social work home visit that received the in-person social work visit | Baseline through 45 days postpartum
  Percentage of women eligible for an in-person social work home visit that received the in-person social work visit
Median number of hospital readmissions - Maternal | Baseline through 365 days postpartum
  Number of hospital readmissions within the first 2 years following delivery
Median number of hospital readmissions - Maternal | Baseline through 730 days postpartum
  Number of hospital readmissions within the first 2 years following delivery
Proportion of women scheduled for a mood check provider visit who received a mood check provider visit | Baseline through 21 days postpartum
  Number of women scheduled for a mood check visit and attended their mood check visit within 21 days of discharge after delivery
Proportion of infants that received recommended immunizations | Baseline through Day 274
  Percentage of infants that received 3 hepatitis B, 2-3 rotavirus (depending on which one is given), 3 diphtheria/tetanus/pertussis, 3 haemophilus influenzae type B, 3 pneumococcal conjugate vaccines, 3 inactivated polio, and 1 flu vaccine within the first 9 months after discharge
Proportion of infants exclusively receiving breastmilk at nurse encounter | Baseline through Day 21
  Percentage of infants exclusively breastfeeding at the time of the nurse home visit within the first 3 weeks after discharge.
Proportion of infants receiving any amount of breastmilk at nurse encounter | Baseline through Day 21
  Percentage of infants receiving any breastmilk at the time of the nurse home visit within the first 3 weeks after discharge
Median number of hospital readmissions - Infant | Baseline through day 365
  Number of hospital readmissions within the first 2 years following discharge.
Median number of hospital readmissions - Infant | Baseline through day 730
  Number of hospital readmissions within the first 2 years following discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth T. Jensen, MPH PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No